CLINICAL TRIAL: NCT04150991
Title: Profiling of the Gut Microbiome in Children With Prader-Willi Syndrome: a Fiber Intervention to Target Hyperphagia (AIM 2)
Brief Title: Fiber Intervention on Gut Microbiota in Children With Prader-Willi Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00069477
Record Dates: First submitted 2019-10-15; First posted 2019-11-05 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Prader-Willi Syndrome; Hyperphagia
Keywords: Fiber; Gut microbiome; Hyperphagia; Prader-Willi Syndrome
MeSH Terms: conditions — Prader-Willi Syndrome; Hyperphagia

STUDY DESIGN:
Intervention Model Description: Participants will receive 3-week fiber/placebo treatment and 3-week alternate fiber/placebo treatment with a 4-week washout period in between.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fiber intervention (Experimental): The investigator's targeted supplemental fiber mixture (35 g total) will be composed of 6g of fiber from oligofructose + 10g from resistant maltodextrin + 12g from acacia gum + 4g from whole foods + 3g from RS2; and will be split into three meals each day.
  Interventions: Other: Fiber intervention
- Placebo treatment (Placebo Comparator): Maltodextrin will be used as a placebo control, as it is digested in the small intestine and thus does not exert local effects in the colon.
  Interventions: Other: Placebo treatment

INTERVENTIONS:
Other: Fiber intervention — Each subject will supplement his/her normal dietary intake with 35 grams of dietary fiber daily for three consecutive weeks.
  Arms: Fiber intervention
Other: Placebo treatment — Each subject will supplement his/her normal dietary intake with an 18.53-g maltodextrin placebo daily for three consecutive weeks.
  Arms: Placebo treatment

SUMMARY:
Prader-Willi syndrome (PWS) is the most common syndromic cause of obesity. Individuals with PWS characteristically experience excessive weight gain and severe hyperphagia with food compulsivity in early childhood, which often leads to the onset of obesity and metabolic complications. The pathogenesis of hyperphagia and progressive weight gain in PWS is far from being understood, and thus efficacious interventions are still under development. Emerging evidence indicates an important etiological contribution of dysbiotic gut microbiota in the hyperphagia, obesity and metabolic abnormalities associated with PWS, implicating a potentially effective target for appetite control and alleviation of obesity in PWS. This study aims to evaluate whether dietary fibers can improve hyperphagia and metabolic profile in children with PWS, and further will determine if these improvements correlate with dietary-fiber-induced changes of the gut microbiota. Twenty children with PWS (age 5-17 years) will receive 3-week fiber or placebo treatment and 3-week alternate treatment with a 4-week washout period in between. A validated PWS-specific hyperphagia questionnaire will be used to assess the severity of hyperphagia in participants. Fasting blood and fecal samples will be collected for the analyses of appetite-related hormones, metabolic biomarkers, bacterial composition and gut metabolites. This study should provide potential new approaches for effective non-pharmacologic treatment of excessive weight gain and hyperphagia associated with PWS to improve overall health and quality of life in affected patients.

DETAILED DESCRIPTION:
Background: Prader-Willi syndrome (PWS) is the most common syndromic cause of obesity. Individuals with PWS characteristically experience excessive weight gain and severe hyperphagia with food compulsivity in early childhood, which often leads to the development of obesity and metabolic complications. The pathogenesis of hyperphagia and progressive weight gain in PWS is far from being understood, and thus efficacious interventions are still being developed. Emerging evidence indicates an important etiological contribution of dysbiotic gut microbiota to the hyperphagia, obesity and metabolic abnormalities associated with PWS, implicating a potentially effective target for appetite control and alleviation of obesity in PWS. The therapeutic potential of manipulating gut microbiota through diet has been scarcely assessed in PWS; more comprehensive evaluations are greatly needed.

Specific objectives: 1) to assess the effects of a 3-week dietary fiber intervention on gut microbiota, hyperphagia, and metabolic profile in children with PWS; 2) to determine whether changes in gut microbial composition and function correlate with changes in the degree of hyperphagia, metabolic hormones, insulin sensitivity, inflammatory markers, and metabolites implicated in cardiometabolic diseases.

Methodological Approach: In a cross-sectional design, 20 children with PWS aged 5 to 17 years will be recruited from the Stollery Children's Hospital, Edmonton. Eligible participants will have normal values of free thyroxine and thyroid-stimulating hormone (either endogenous or with thyroxine replacement) as well as stable body weight and growth hormone dose. Children with other clinically significant disease (diabetes mellitus, chronic inflammatory bowel disease, chronic severe liver or kidney disease), or recent use of medications known to affect body weight and gut microbiota (investigational drugs, antibiotics, prebiotic and/or probiotic supplements) will be excluded. Participants will be randomly assigned to consume either 35 g supplemental fiber mixture/d (oligofructose, resistant maltodextrin, acacia gum, whole foods, and resistant starch type II) or an equicaloric dose of a 17.6-g maltodextrin placebo/d (GLOBE® Plus 10 DE Maltodextrin 100200; Ingredion) for 3 wk. This will be followed by a 4-wk washout period and an alternate treatment for another 3 wk. Fecal samples will be collected to analyze gut microbiota composition (using 16S ribosomal ribonucleic acid [rRNA] tag sequencing) and function (metabolites produced by microbiota: SCFAs and bile acids). Microbiota composition will be characterized at phylum to genus level, and sequences will be clustered to Operational Taxonomic Units to calculate alpha-diversity (by Shannon index). Fasting blood samples will be used to measure appetite-related hormones, and metabolic and inflammatory markers. A validated PWS-specific hyperphagia questionnaire will be used to assess participants' food-related behaviors. A 3-day dietary record including physical activity questions will be administered for the assessment of macro- and-micronutrient intake and diet quality as well as physical activity level of the participants. In addition, anthropometric data (body weight, height and waist circumference [WC]) will be obtained to track changes.

Outcomes: 1) Primary outcome: Change in hyperphagia score; 2) Secondary outcomes: Changes in: a. Fecal microbial composition and function; b. Hormones (acylated ghrelin, PYY, GLP-1, adiponectin and leptin; c. Metabolic and inflammatory markers (glucose, insulin, lipids, AST, ALT, hs-CRP); d. Metabolomics profile (amino acids, branched chain keto acids, acylcarnitines, ceramides, TMAO, choline and betaine); and e. body weight, height and WC.

Deliverables: 1) the feasibility of using a fiber intervention to reduce hyperphagia and improve metabolism and inflammation via beneficial changes in the microbiota in children with PWS; 2) the particular microbial composition and functional profiles associated with metabolic improvement and/or weight loss can aid in the future development of microbial-targeted prebiotic therapies. Results from this study will be used to guide the design of effective treatment strategies to reduce hyperphagia and improve metabolic health in children with PWS.

ELIGIBILITY:
Inclusion Criteria:

* PWS diagnosis confirmed by chromosome analysis;
* Age 5-25 years;
* Informed consent/ assent and willingness to comply with study procedures;
* Free T4, TSH values in the normal range (either endogenous or with thyroxine replacement);
* Weight stable (Body Mass Index [BMI] percentile fluctuation < 5%) over the preceding 2 months;
* Stable growth hormone dose over the prior 6 months.

Exclusion Criteria:

* Other clinically significant diseases including diabetes mellitus, chronic inflammatory bowel disease, chronic severe liver, kidney disease or neurologic disorders;
* Concomitant use of medication/investigational drug known to affect body weight in the past year;
* Antibiotic use in the past 60 days;
* Probiotic and/or prebiotic supplements use in the past 30 days.

Ages: 5 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2023-02-22 (Actual); Study Completion 2023-02-22 (Actual)

PRIMARY OUTCOMES:
Changes in hyperphagia | Week 1, 3, 7 &10
  Change in hyperphagia will be measured by the Hyperphagia Questionnaire for Clinical Trials. This questionnaire consists of nine items with responses ranging from 0-4 units each (possible total score range: 0-36; higher scores indicate higher degree of hyperphagia; reductions in score from baseline indicate improvement in hyperphagia-related behaviors).

SECONDARY OUTCOMES:
Changes in gut microbiota | Week 1, 3, 7 &10
  16SrRNA-sequencing and whole metagenome sequencing will performed to determine gut microbial community changes induced by dietary fibers.
Changes in appetite and satiety hormones | Week 1, 3, 7 &10
  Fasting blood samples will be collected to quantify the plasma concentrations of circulating appetite regulating hormones.
Changes in inflammatory status | Week 1, 3, 7 &10
  Plasma levels of C-Reactive Protein (mg/L) will be measured to determine if fiber intervention can improve inflammatory outcomes.
Changes in metabolic markers | Week 1, 3, 7 &10
  Plasma levels of metabolic markers will be measured determine if fiber intervention can improve metabolic functions.
Changes in metabolomics | Week 1, 3, 7 &10
  Plasma levels of metabolomics will be measured determine if fiber intervention can improve metabolic functions.
Change in anthropometric measurements | Week 1, 3, 7 &10
  Weight will be measured to the nearest 0.1kg using a calibrated scale. Height will be measured to the nearest 0.1cm using a wall-mounted stadiometer. Waist circumference will be measured to the nearest 0.1 cm at the top of the iliac crest using an inelastic measuring tape. Weight and height will be combined to report BMI in kg/m^2.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Haqq, MD, MHS, Principal Investigator — University of Alberta
Locations (1):
- Li Ka Shing Centre for Health Research Innovation, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Irizarry KA, Miller M, Freemark M, Haqq AM. Prader Willi Syndrome: Genetics, Metabolomics, Hormonal Function, and New Approaches to Therapy. Adv Pediatr. 2016 Aug;63(1):47-77. doi: 10.1016/j.yapd.2016.04.005. No abstract available. PMID 27426895
- [Background] Irizarry KA, Bain J, Butler MG, Ilkayeva O, Muehlbauer M, Haqq AM, Freemark M. Metabolic profiling in Prader-Willi syndrome and nonsyndromic obesity: sex differences and the role of growth hormone. Clin Endocrinol (Oxf). 2015 Dec;83(6):797-805. doi: 10.1111/cen.12766. Epub 2015 Apr 1. PMID 25736874
- [Background] Zhang C, Yin A, Li H, Wang R, Wu G, Shen J, Zhang M, Wang L, Hou Y, Ouyang H, Zhang Y, Zheng Y, Wang J, Lv X, Wang Y, Zhang F, Zeng B, Li W, Yan F, Zhao Y, Pang X, Zhang X, Fu H, Chen F, Zhao N, Hamaker BR, Bridgewater LC, Weinkove D, Clement K, Dore J, Holmes E, Xiao H, Zhao G, Yang S, Bork P, Nicholson JK, Wei H, Tang H, Zhang X, Zhao L. Dietary Modulation of Gut Microbiota Contributes to Alleviation of Both Genetic and Simple Obesity in Children. EBioMedicine. 2015 Jul 10;2(8):968-84. doi: 10.1016/j.ebiom.2015.07.007. eCollection 2015 Aug. PMID 26425705